CLINICAL TRIAL: NCT02093117
Title: Effect of an Alveolar Recruitment Maneuver on Subdural Pressure, Brain Swelling and Cerebral Perfusion Pressure in Patients Undergoing Supratentorial Tumour Resection
Brief Title: Neurosurgery Recruitment Maneuver Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Alana Flexman, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H14-00009
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2015-12

CONDITIONS: Subdural Pressure During Supratentorial Brain Tumour Resection
Keywords: Supratentorial neurosurgery; Recruitment maneuver; Subdural pressure; Brain relaxation; Cerebral perfusion pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recruitment maneuver (Experimental): The recruitment maneuver will involve application of continuous positive airway pressure of 30 cm of water for 30 seconds.
  Interventions: Procedure: Recruitment maneuver
- Sham recruitment maneuver (Sham Comparator): The sham recruitment maneuver will involve application of continuous positive airway pressure of 5 cm of water for 30 seconds.
  Interventions: Procedure: Sham recruitment maneuver

INTERVENTIONS:
Procedure: Recruitment maneuver — continuous positive airway pressure of 30 cm of water for 30 seconds
  Arms: Recruitment maneuver
Procedure: Sham recruitment maneuver — Continuous positive airway pressure of 5 cm of water for 30 seconds
  Arms: Sham recruitment maneuver

SUMMARY:
Background. Patients undergoing neurosurgical procedures experience higher rates of postoperative respiratory failure compared to the broader surgical population. Lung-protective ventilation strategies, including alveolar recruitment maneuvers may be beneficial. Despite this potential benefit, the effect of high levels of continuous airway pressure on intracranial pressure, brain swelling and cerebral perfusion must be defined prior to applying this intervention to the neurosurgical population.

Objectives. The primary objective is to determine the effect of an alveolar recruitment maneuver on subdural pressure in patients undergoing supratentorial tumour resection. The secondary objectives are to determine the effect of an alveolar recruitment maneuver on 1) brain bulk score and 2) cerebral perfusion pressure in patients undergoing supratentorial tumour resection.

Hypothesis. The investigators hypothesize that an alveolar recruitment maneuver of 30 cm of water over 30 seconds will not result in a clinically-important (>3 mmHg) increase in subdural pressure.

Methods. This single center, randomized, cross-over study will enroll 30 American Society of Anesthesiologists Classification I-III patients scheduled to undergo supratentorial brain tumour resection at Vancouver General Hospital. All patients will receive a standardized general anesthetic including invasive blood pressure monitoring. After removal of the bone flap, subdural pressure will be measured using a sterile 22-gauge plastic cannula. Brain bulk will be assessed using a validated 4-point scale. After baseline arterial and subdural pressure determination and brain swelling assessments, patients will be randomized to receive either a recruitment maneuver of 30 cm of water for 30 seconds or a sham recruitment maneuver of 5 cm of water for 30 seconds. Maximal subdural pressure and minimum mean arterial pressure during the maneuver will be noted, and the neurosurgeon will be asked to score the brain bulk. After a 2-minute equilibration period, the protocol will be repeated with the alternate group allocation.

Statistical Analysis. Our sample size calculation, based on our primary outcome (subdural pressure), determined that a sample size of 22 patients would allow us to detect a difference of 3.5 mmHg in subdural pressure assuming a type I error of 0.05, a type II error of 0.2 and two-sided significance testing. The subdural pressure during the recruitment maneuver as compared to the sham maneuver will be analyzed using a paired t-test. The brain bulk score will be compared using a Wilcoxon signed rank test. All data analysis will be performed with STATA 12.1 (StataCorp, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years of age) scheduled for craniotomy for resection of a supratentorial brain tumour who are American Society of Anesthesiologist's class I to III are eligible to participate.

Exclusion Criteria:

* Patient with altered level of consciousness or unstable/deteriorating neurologic status preoperatively will be excluded.
* In addition, if the neurosurgeon considers the mass effect too great to safely participate the patient will be excluded. Baseline subdural pressure will be measured prior to randomization
* Patients with a subdural pressure greater than 20 mmHg will be excluded.
* Other exclusion criteria include significant cardiac disease (e.g. ejection fraction < 40 percent, significant valvular disease, pulmonary hypertension), sepsis, hypovolemia and prior lung resection or history of pneumothorax.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Subdural pressure | At baseline and within 30 seconds of recruitment maneuver or sham
  Change in subdural pressure (mmHg) during a recruitment maneuver as compared to a sham recruitment maneuver

SECONDARY OUTCOMES:
Brain relaxation score | At baseline and within 30 seconds of recruitment maneuver or sham
  Change in surgeon-assessed brain relaxation score (1-4) at the end of the recruitment maneuver as compared to the sham recruitment maneuver
Cerebral perfusion pressure | At baseline and within 30 seconds of recruitment maneuver or sham
  Change in cerebral perfusion pressure at the end of the recruitment maneuver as compared to the sham recruitment maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Alana Flexman, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Flexman AM, Gooderham PA, Griesdale DE, Argue R, Toyota B. Effects of an alveolar recruitment maneuver on subdural pressure, brain swelling, and mean arterial pressure in patients undergoing supratentorial tumour resection: a randomized crossover study. Can J Anaesth. 2017 Jun;64(6):626-633. doi: 10.1007/s12630-017-0863-7. Epub 2017 Mar 24. PMID 28342045